CLINICAL TRIAL: NCT02393781
Title: Adrenomedullin and Outcome in Severe Sepsis and Septic Shock. The AdrenOSS Study.
Brief Title: Adrenomedullin and Outcome in Severe Sepsis and Septic Shock
Acronym: AdrenOSS
Status: Completed | Type: Observational
Sponsor: Sphingotec GmbH (Industry)
Collaborators: Fondation Transplantation_EDDH (Unknown); Hopital Lariboisière (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A01906-41
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: severe sepsis; septic shock; adrenomedullin; organ dysfunction
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples without DNA Blood samples (heparin-, EDTA-, EDTA/aprotinin plasma) and urine samples will be collected at the admission, day 2, day 3 and the day of discharge for measuring ADM and other markers
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this prospective study is to assess the prognostic value of bioactive plasma adrenomedullin (ADM) in 600 patients with severe sepsis or septic shock in an international multicenter study and to validate the findings concerning the association of ADM concentration and the use of vasopressor therapy, organ failure and outcome.

DETAILED DESCRIPTION:
Sepsis involves an overactive inflammatory response to severe bacterial infection that can compromise vascular integrity and cause tissue edema, organ dysfunction and death. Adrenomedullin (ADM) has attracted the interest of researchers because of its powerful physiological functions. An anti-ADM antibody reduced the norepinephrine infusion rates required to achieve hemodynamic targets, increased urine flow and improved creatinine clearance, which ultimately resulted in attenuated systemic inflammation and tissue apoptosis, during resuscitated cecal ligation and puncture (CLP)-induced septic shock in mice.

In humans, plasma ADM has been determined only in a small number of sepsis patients, and - except from one study - the assays used did not selectively measure the bioactive ADM form and have been considered not reliable. Therefore, the potential value of determining plasma ADM in such patients cannot yet be ascertained and the optimal cut off needs to be validated in future studies

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients admitted in intensive care unit for severe sepsis or septic shock according to international, standardized criteria,transferred from another intensive care unit less than 24 hours after the primary admission, or being treated with vasopressors for less than 24 hours in the prior ICU
* Signed Consent form

Exclusion Criteria:

* Age < 18 years
* Severe sepsis or septic shock patients transferred from another intensive care unit later than 24 hours after the primary admission or being treated with vasopressors for more than 24 hours in the prior ICU
* Pregnant women
* Vegetative coma
* Participation in an interventional clinical trial in the preceding month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 patients admitted in intensive care unit of 26 hospitals, in 5 countries, with diagnosis of severe sepsis or septic shock, will be included in this study.
Sampling Method: Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
rate of all-cause mortality | Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Mebazaa, Pr, Principal Investigator — Hôpital Lariboisière, France; Pierre François Laterre, Pr, Principal Investigator — Clinique Universitaire St Luc, Belgique
Locations (24):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - CH Jolimont, La Louvière
  - Clinique St Pierre, Ottignies
- France (12):
  - Centre Hospitalier d'Angers, Angers
  - Centre Hospitalier d'Angoulême, Angoulême
  - Hopital Estaing, Clermont-Ferrand
  - Hôpital Louis Mourier,, Colombes
  - CHD de la Vendée, La Roche-sur-Yon
  - CHU Dupuytren, Limoges
  - Hôpital St Louis, Paris
  - Hôpital Bichat Claude-Bernard, Paris
  - Hôpital Lariboisière, Paris
  - Nouvel Hôpital Civil, Strasbourg
  - Hôpital de Hautepierre, Strasbourg
  - CHRU Tours, Tours
- Germany (5):
  - Klinik für Operative Intensivmedizin und Intermediate Care, Aachen
  - Klinikum Augsburg, Augsburg
  - Klinik für Anästhesiologie und Operative Intensivmedizin, Universitätsklinikum Köln, Cologne
  - Klinik für Anästhesie, Intensivmedizin und Schmerztherapie, HELIOS-Klinikum Erfurt,, Erfurt
  - Universitätsklinikum Jena, Jena
- Italy (2):
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Policlinico Universitario A. Gemelli, Roma
- Netherlands (2):
  - Medisch Spectrum Twente; Departement of Intensive Care, Enschede, Enschede
  - UMC Radboudziekenhuis, Dept. Intensive Care, Nijmegen

REFERENCES:
- [Derived] Jolly L, Carrasco K, Salcedo-Magguilli M, Garaud JJ, Lambden S, van der Poll T, Mebazaa A, Laterre PF, Gibot S, Boufenzer A, Derive M. sTREM-1 is a specific biomarker of TREM-1 pathway activation. Cell Mol Immunol. 2021 Aug;18(8):2054-2056. doi: 10.1038/s41423-021-00733-5. Epub 2021 Jul 19. No abstract available. PMID 34282296
- [Derived] Blet A, Deniau B, Santos K, van Lier DPT, Azibani F, Wittebole X, Chousterman BG, Gayat E, Hartmann O, Struck J, Bergmann A, Antonelli M, Beishuizen A, Constantin JM, Damoisel C, Deye N, Di Somma S, Dugernier T, Francois B, Gaudry S, Huberlant V, Lascarrou JB, Marx G, Mercier E, Oueslati H, Pickkers P, Sonneville R, Legrand M, Laterre PF, Mebazaa A; AdrenOSS-1 Study Investigators. Monitoring circulating dipeptidyl peptidase 3 (DPP3) predicts improvement of organ failure and survival in sepsis: a prospective observational multinational study. Crit Care. 2021 Feb 15;25(1):61. doi: 10.1186/s13054-021-03471-2. PMID 33588925
- [Derived] Mebazaa A, Geven C, Hollinger A, Wittebole X, Chousterman BG, Blet A, Gayat E, Hartmann O, Scigalla P, Struck J, Bergmann A, Antonelli M, Beishuizen A, Constantin JM, Damoisel C, Deye N, Di Somma S, Dugernier T, Francois B, Gaudry S, Huberlant V, Lascarrou JB, Marx G, Mercier E, Oueslati H, Pickkers P, Sonneville R, Legrand M, Laterre PF; AdrenOSS-1 study investigators. Circulating adrenomedullin estimates survival and reversibility of organ failure in sepsis: the prospective observational multinational Adrenomedullin and Outcome in Sepsis and Septic Shock-1 (AdrenOSS-1) study. Crit Care. 2018 Dec 21;22(1):354. doi: 10.1186/s13054-018-2243-2. PMID 30583748
- [Derived] Hollinger A, Wittebole X, Francois B, Pickkers P, Antonelli M, Gayat E, Chousterman BG, Lascarrou JB, Dugernier T, Di Somma S, Struck J, Bergmann A, Beishuizen A, Constantin JM, Damoisel C, Deye N, Gaudry S, Huberlant V, Marx G, Mercier E, Oueslati H, Hartmann O, Sonneville R, Laterre PF, Mebazaa A, Legrand M. Proenkephalin A 119-159 (Penkid) Is an Early Biomarker of Septic Acute Kidney Injury: The Kidney in Sepsis and Septic Shock (Kid-SSS) Study. Kidney Int Rep. 2018 Aug 22;3(6):1424-1433. doi: 10.1016/j.ekir.2018.08.006. eCollection 2018 Nov. PMID 30450469